CLINICAL TRIAL: NCT01529242
Title: A Double-blind, Randomized, Multicenter Parallel-group Study on Efficacy of Desloratadine and Prednisolone Association Compared to Dexchlorpheniramine and Betamethasone Association in Children (2-12 Years) With Acute Cutaneous Rash
Brief Title: Comparison of Desloratadine Associated With Prednisolone Oral Solution Versus Dexchlorpheniramine Associated With Betamethasone for Cutaneous Rash Treatment
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: By sponsor decision due to difficulty of recruitment
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DPUEMS1111
Record Dates: First submitted 2012-02-06; First posted 2012-02-08 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Cutaneous Hypersensitivity
MeSH Terms: interventions — desloratadine; Prednisolone; dexchlorpheniramine; Betamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desloratadine + Prednisolone (Experimental): desloratadine 0,5 mg/ml + prednisolone 4 mg/ml - oral solution
  Interventions: Drug: Desloratadine + Prednisolone
- Dexchlorpheniramine + Betamethasone (Active Comparator): dexchlorpheniramine maleate 0,4 mg/ml + Betamethasone 0,05 mg/ml - oral solution
  Interventions: Drug: Dexchlorpheniramine + Betamethasone

INTERVENTIONS:
Drug: Desloratadine + Prednisolone — Children (2 to 5 years): 2.5 ml 3 times a day Children (6 to 12 years): 5.0 ml 3 times a day
  Arms: Desloratadine + Prednisolone
Drug: Dexchlorpheniramine + Betamethasone — Children (2 to 5 years): 2.5 ml 3 times a day Children (6 to 12 years): 5.0 ml 3 times a day
  Arms: Dexchlorpheniramine + Betamethasone

SUMMARY:
The purpose of this study is to evaluate the non-inferiority clinical efficacy of two different drug associations in the treatment of acute cutaneous rash in children between 2 and 12 years old.

DETAILED DESCRIPTION:
* double-blind, non-inferiority, prospective, parallel group trial.
* Experiment duration: 05 days.
* 03 visits (day 0, 48 hours and day 5).
* Efficacy will be evaluated for acute cutaneous rash based on symptoms score
* Adverse events evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Consent of the patient or legal guardian;
* Clinical diagnosis of acute cutaneous rash defined by the presence of erythematous papules on healthy skin, different sizes, itchy and fleeting
* Children aged between 2 and 11 years and 11 months (up to 30 kg);

Exclusion Criteria:

* Participation in clinical trial in 30 days prior to study entry;
* Patients with history of hypersensitivity to desloratadine or prednisolone or with corticosteroids use contraindications ;
* Patients with any clinically significant disease other than cutaneous rash including hematopoietic, cardiovascular, renal, neurological, psychiatric or autoimmune disorders;
* Patients on treatment with monoamine oxidase inhibitors (MAOIs);
* Patients diagnosed with other dermatoses

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-10-20 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment in acute cutaneous rash based on symptoms score | 5 days
  The differences in the intensity of signs and symptoms of acute cutaneous rash between the beginning and end of the study will be used as the primary endpoint of clinical efficacy
  .

SECONDARY OUTCOMES:
Safety will be evaluated by the adverse event occurrences | 5 days
  Adverse events will be recorded and followed in order to evaluate safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Dirceu Solé, MD, Principal Investigator — Federal University of São Paulo
Locations (3):
- Brazil (3):
  - Allergisa, Campinas, São Paulo
  - Alergoalpha, São Paulo, São Paulo
  - Hospital Nipo Brasileiro, São Paulo, São Paulo